CLINICAL TRIAL: NCT04170465
Title: Investigation of the Potential Beneficial Effect of Adding Metformin to Neoadjuvant Chemotherapy in Patients With Breast Cancer (METNEO)
Brief Title: Role of Adding Metformin to Neoadjuvant Chemotherapy in Patients With Breast Cancer (METNEO)
Acronym: METNEO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Damanhour University (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 919PP18
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer Female
Keywords: Metformin; locally advanced breast cancer; neoadjuvant
MeSH Terms: interventions — Metformin; Doxorubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin group (Experimental): Patients will receive AC-T neoadjuvant chemotherapy in addition to oral metformin HCl (850 mg tablets, twice per day, for 6 months) (n= 30)
  Interventions: Drug: Metformin Hydrochloride 850 mg Tablets; Drug: AC-T chemotherapy regimen
- Control group (Active Comparator): Patients will receive AC-T neoadjuvant chemotherapy alone (n= 30)
  Interventions: Drug: AC-T chemotherapy regimen

INTERVENTIONS:
Drug: Metformin Hydrochloride 850 mg Tablets — Oral administration of Metformin hydrochloride 850 mg tablets (1700 mg/day) daily until the completion of neoadjuvant chemotherapy cycles
  Other Names: Cidophage 850 mg
  Arms: Metformin group
Drug: AC-T chemotherapy regimen — AC: (Doxorubicin 60 mg/m2 IV + cyclophosphamide 600 mg/m2 IV) for 4 cycles every 3 weeks followed by Taxol cycles (Paclitaxel 80 mg/m2 IV) once weekly for 12 weeks.
  Other Names: AC (doxorubicin [Adriamycin] + cyclophosphamide) followed by paclitaxel (Taxol)

SUMMARY:
Metformin, the widely prescribed oral hypoglycemic drug, is well known for its established efficacy, favorable safety profile, and low cost. Metformin has recently received increasing attention because of its potential antitumorigenic effects that are thought to be independent of its hypoglycemic effects. It has been extensively studied in preclinical models, which have implicated several molecular pathways in its antitumor activity.

Metformin was proved to have anti-proliferative and apoptotic effects on tumor cells.Moreover, metformin enhances the T-cell mediated immune response to tumor tissue and fights metastases. Also, epidemiological studies have shown that metformin, but not other antidiabetic drugs, reduces cancer incidence and improves survivability in diabetic cancer patients.

The proposed research in this application will investigate two prime questions with regards to the combined use of metformin together with traditional neoadjuvant chemotherapy in breast cancer patients. First, the hypothesis that the simultaneous use of metformin along with doxorubicin/cyclophosphamide/paclitaxel neoadjuvant protocol produces better antitumor outcomes will be tested. Second, the study will examine if the improved apoptotic effect of such regimen is paralleled by exaggerated stimulatory influences on apoptosis biomarkers.

DETAILED DESCRIPTION:
1. Ethical committee approval will be obtained from Ethics committee of Faculty of Pharmacy, Damanhour University.
2. All participants should agree to take part in this clinical study and will provide informed consent.
3. Sixty female breast cancer patients, who are candidates for neoadjuvant chemotherapy, will be recruited from the Medical Research Institute, Oncology department, Alexandria University, Alexandria.
4. The 60 participants will be randomly assigned into 2 arms:

   * Control arm (n=30): will be treated with AC-Taxol regimen (AC: Doxorubicin 60 mg/m2 IV + cyclophosphamide 600 mg/m2 IV) for 4 cycles every 3 weeks. Subsequent Taxol cycles (Paclitaxel 80mg/m2 IV) once weekly for 12 weeks.
   * Metformin arm (n=30): will be treated with the AC-Taxol regimen mentioned above together with Metformin 850 mg tablets orally twice per day (1700 mg/day).
5. All patients will be submitted to:

   * Full patient history and clinical examination.
   * Routine follow up before each chemotherapy cycle (complete blood picture, liver function tests, renal function tests).
   * Routine Echocardiography before each chemotherapy cycle.
6. All patients will be monitored for the incidence of chemotherapy toxicities during neoadjuvant therapy.
7. After completion of the neoadjuvant therapy, participants will undergo surgical tumor removal. The excised tumor will be collected, and the expression of apoptosis biomarkers and the pathologic complete response (pCR) will be assessed.
8. Patients demographic data will be recorded with respect to age, weight and disease history.
9. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.
10. Results, conclusion, discussion and recommendations will be given.

ELIGIBILITY:
Inclusion Criteria:

1. Females ≥ 18 years of age and < 65 years.
2. Unilateral or bilateral primary carcinoma of the breast confirmed.
3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-2.
4. Clinically measurable tumor size who are candidates for neoadjuvant therapy.
5. No evidence of distant metastasis.
6. Normal renal and liver functions.
7. Non-diabetics.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Prior cancer chemotherapy.
3. Heart disease or reduced cardiac output with left ventricular ejection fraction < 50%.
4. Metastatic breast cancer patients.
5. Patients with hepatic impairment.
6. Patients with renal impairment.
7. Diabetics.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect on tumor apoptosis | 6 months
  Tissue level of the apoptosis biomarker in the excised tumor.
Chemotherapy toxicities | 6 months
  Monitoring the incidence of chemotherapy toxicities during neoadjuvant therapy

SECONDARY OUTCOMES:
Pathologic complete response rate (pCR) | 6 months
  Pathologic complete response rate defined as the absence of residual invasive cancer in the resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M El-Mas, PhD, Study Director — Professor in Pharmacology, Faculty of Pharmacy, Alexandria University; Yasser M El-Kerm, PhD, Study Director — Professor in Clinical Oncology, Medical Research Institute,Alexandria University; Maged W Helmy, PhD, Study Chair — Professor in Pharmacology, Faculty of pharmacy, Damanhour University; Amira B Kassem, PhD, Study Chair — Lecturer in Clinical Pharmacy, Faculty of Pharmacy, Damanhour University; Noha A El-Bassiouny, PhD, Study Chair — Lecturer in Clinical Pharmacy, Faculty of Pharmacy, Damanhour University; Manar A Serageldin, Bachelor, Principal Investigator — Teaching assistant in Pharmacology, Faculty of Pharmacy, Alexandria University
Locations (1):
- Damanhour University, Beheira, Egypt

IPD SHARING:
Plan to Share IPD: No
Summary of all relevant data will be shared

REFERENCES:
- [Derived] Serageldin MA, El-Bassiouny NA, El-Kerm Y, Aly RG, Helmy MW, El-Mas MM, Kassem AB. A randomized controlled study of neoadjuvant metformin with chemotherapy in nondiabetic breast cancer women: The METNEO study. Br J Clin Pharmacol. 2024 Dec;90(12):3160-3175. doi: 10.1111/bcp.16193. Epub 2024 Aug 7. PMID 39113190
- [Derived] Serageldin MA, Kassem AB, El-Kerm Y, Helmy MW, El-Mas MM, El-Bassiouny NA. The Effect of Metformin on Chemotherapy-Induced Toxicities in Non-diabetic Breast Cancer Patients: A Randomised Controlled Study. Drug Saf. 2023 Jun;46(6):587-599. doi: 10.1007/s40264-023-01305-4. Epub 2023 May 2. PMID 37131014